CLINICAL TRIAL: NCT01423487
Title: Efficacy and Safety of Metformin in Preventing Patients With Risperidone From Weight Gain and Amenorrhea:a 24-week, Randomized, Placebo-controlled, Double-blind, Fixed-dose Study
Brief Title: Efficacy and Safety of Metformin in Preventing Patients With Risperidone From Weight Gain and Amenorrhea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to obtain informed consent
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jing-Ping Zhao, Professor,Deputy Director of Mental Health Institute of The Second Xiangya Hospital, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSUXXEYYJYS-051
Record Dates: First submitted 2011-08-18; First posted 2011-08-26 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Weight Gain; Amenorrhea
Keywords: Metformin; Risperidone; Prevention; weight gain; Amenorrhea
MeSH Terms: conditions — Weight Gain; Amenorrhea | interventions — Metformin; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- efficacy and safety (Experimental): To investigate the efficacy and safety of Metformin in preventing patients with Risperidone from weight gain and amenorrhea.
  Interventions: Drug: Metformin
- placebo comparator (Placebo Comparator): To investigate whether plcebo also could preventing patients with Risperidone from weight gain and amenorrhea.
  Interventions: Other: Starch tablets

INTERVENTIONS:
Drug: Metformin — 0.5g bid 26 weeks
  Arms: efficacy and safety
Other: Starch tablets — 0.5g bid 26 weeks
  Arms: placebo comparator

SUMMARY:
Some previous studies has demonstrated that Metformin can improve the weight gain which caused by antipsychotics. An our study, which will be published, also found that Metformin can improve the amenorrhea for patients with antipsychotics, approximately 60% patients recovery period. So the present study was designed to investigate the efficacy and safety of Metformin in preventing patients with Risperidone from weight gain and amenorrhea.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-40 years.
2. diagnosis of schizophrenia (naive first-episode) as defined in DSM-IV axis I.
3. At screening, patients were required to have total score ≥60 on Positive and Negative Syndrome Scale (PANSS) and ≥4 on the Clinical Global Impression-severity scale (CGI-S).
4. treat with Risperidone.
5. Never participate in a diet control nor in other weight loss programs, and have a normal Period.
6. Written informed consents could be obtained from patients(or their Legal guardian).

Exclusion Criteria:

1. Female patients, those who were in the period of pregnancy and lactation, or plan pregnancy, were excluded.
2. Patients with serious physical disease patients, just like Epilepsy, liver and kidney dysfunction, diabetes, blood diseases, etc were excluded.
3. At screening, patients with abnormal results in physical examination, laboratory test, or electrocardiogram (ECG) were excluded.
4. Patients were also excluded if they met primary DSM-IV axis I psychiatric disorders other than schizophrenia, or ever used psychoactive substance.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in weight at 24 weeks | baseline, 8 week, 16 week, 24 week
  The data will be presented

SECONDARY OUTCOMES:
Change from Baseline in menstruation at 24 weeks | baseline, 4 week, 8 week, 12 week, 16 week, 20 week, 24 week
  The data will be presented

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Ping Zhao, Dr., Ph.D., Study Chair — Mental Health Institute of The Second Xiangya Hospital, Central South University
Locations (1):
- Mental Health Institute of The Second Xiangya Hospital, Changsha, Hunan, China

REFERENCES:
- [Background] Wu RR, Zhao JP, Jin H, Shao P, Fang MS, Guo XF, He YQ, Liu YJ, Chen JD, Li LH. Lifestyle intervention and metformin for treatment of antipsychotic-induced weight gain: a randomized controlled trial. JAMA. 2008 Jan 9;299(2):185-93. doi: 10.1001/jama.2007.56-b. PMID 18182600